CLINICAL TRIAL: NCT05946031
Title: Testing the Experimental Tobacco Marketplace: Examination and Comparison of Different Methods
Brief Title: Testing the ETM: Examination and Comparison of Different Methods
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #24-837
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-12

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Participants will complete two Experimental Marketplace conditions, representing one with real and one with hypothetical purchasing outcomes. Within each condition, taxes will be increased proportionally across 6 trials to examine how cigarette purchasing, substitution, and poly-tobacco purchasing (i.e., diversity in products purchased) are affected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-lab procedures (Experimental): Exclusive cigarette smokers will be recruited and will experience all study procedures in the laboratory.
  Interventions: Drug: Reat ETM; Drug: Hypothetical ETM
- Remote procedures (Experimental): Exclusive cigarette smokers will be recruited and will experience all study procedures remotely.
  Interventions: Drug: Reat ETM; Drug: Hypothetical ETM

INTERVENTIONS:
Drug: Reat ETM — Exclusive cigarette smokers will be recruited and will be exposed to the real ETM condition in which tobacco purchases are real and they receive products from one randomly selected trial.
Drug: Hypothetical ETM — Exclusive cigarette smokers will be recruited and will be exposed to the hypothetical ETM condition in which tobacco purchases are hypothetical and they don't receive any products.

SUMMARY:
This study will experimentally assess the comparability of in-lab and remote procedures with hypothetical and real ETM purchase outcomes.

DETAILED DESCRIPTION:
In a between-group within-subject repeated measures design, participants will be randomly assigned to one of two procedures (in-lab or remote; between-group) and complete two conditions (real and hypothetical; within-subject), which include six trials assessing increasing cigarette prices.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Be at least 21 years of age or older
* Stable tobacco use patterns for at least three months
* Smoke at least 5 cigarettes daily
* Use other tobacco products less than weekly
* Have access to a computer and internet

Exclusion Criteria:

* report uncontrolled physical or mental health conditions (e.g., uncontrolled diabetes, high blood pressure, major depressive disorder, etc.),
* use of smoking cessation medications (e.g., nicotine replacement, bupropion, varenicline) in the past 30 days,
* report concrete, immediate plans to alter/quit using their usual tobacco products in the next 30 days,
* be pregnant or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-07-28 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Cigarette demand | 1 day
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Other product prices in the ETM will remain constant. To obtain dependent measures of demand, participants' purchasing of the price-manipulated commodity in the ETM task will be fit to a modified exponential equation to quantify the relationship between the price of each commodity and purchasing: Q=Q0*10k(exp(-αQ0C)-1) where Q is purchasing of the commodity, C is the price, Q0 is the derived initial purchasing without cost constraints (demand intensity), k is the span of the function in logarithmic units, and α is the demand elasticity.
Nicotine/tobacco products substitution | 1 day
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Other product prices in the ETM will remain constant. To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators will use ordinary least squares regression to model the relationship of the price-manipulated product to predict total quantity purchased of the price-constant product.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Freitas-Lemos, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.